CLINICAL TRIAL: NCT02564315
Title: The Long-Term Quitting Study: Testing Relapse Recovery Intervention Components
Brief Title: The Long-Term Quitting (Smoking Cessation) Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Penn State University (Other); University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-1041 LongTermQuitting; A534253 (Other: UW, Madison); SMPH/MEDICINE/GEN INT MD (Other: UW, Madison)
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Smoking Cessation
Keywords: Smoking; Cessation; Tobacco; Relapse
MeSH Terms: conditions — Smoking Cessation; Smoking; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- Reduction/Supportive+Skill Counseling (Active Comparator): This arm includes Phase 2 (Preparation) Reduction Treatment and Phase 3 (Cessation) Supportive Counseling and Skill Training Counseling. More specifically, treatments include the following:
  Phase 2: Nicotine Mini-Lozenge for 11 Months; Preparation Phase Behavioral Reduction Counseling;
  Phase 3: Cessation Phase Supportive Counseling; Cessation Phase Skill Training Counseling; Cessation Phase Nicotine Patch + Nicotine Mini-Lozenge
  Interventions: Drug: Nicotine Mini-Lozenge for 11 Months; Behavioral: Preparation Phase Behavioral Reduction Counseling; Behavioral: Cessation Phase Supportive Counseling; Behavioral: Cessation Phase Skill Training Counseling; Drug: Cessation Phase Nicotine Patch + Nicotine Mini-Lozenge
- Reduction/Supportive Counsel+Brief Info (Active Comparator): This arm includes Phase 2 (Preparation) Reduction Treatment and Phase 3 (Cessation) Supportive Counseling and Brief Information. More specifically, treatments include the following:
  Phase 2: Nicotine Mini-Lozenge for 11 Months; Preparation Phase Behavioral Reduction Counseling;
  Phase 3: Cessation Phase Supportive Counseling; Cessation Phase Brief Information; Cessation Phase Nicotine Patch + Nicotine Mini-Lozenge
  Interventions: Drug: Nicotine Mini-Lozenge for 11 Months; Behavioral: Preparation Phase Behavioral Reduction Counseling; Behavioral: Cessation Phase Supportive Counseling; Behavioral: Cessation Phase Brief Information; Drug: Cessation Phase Nicotine Patch + Nicotine Mini-Lozenge
- Reduction/Skill Counseling+Brief Info (Active Comparator): This arm includes Phase 2 (Preparation) Reduction Treatment and Phase 3 (Cessation) Skill Training Counseling and Brief Information. More specifically, treatments include the following:
  Phase 2: Nicotine Mini-Lozenge for 11 Months; Preparation Phase Behavioral Reduction Counseling;
  Phase 3: Cessation Phase Skill Training Counseling; Cessation Phase Brief Information; Cessation Phase Nicotine Patch + Nicotine Mini-Lozenge
  Interventions: Drug: Nicotine Mini-Lozenge for 11 Months; Behavioral: Preparation Phase Behavioral Reduction Counseling; Behavioral: Cessation Phase Skill Training Counseling; Behavioral: Cessation Phase Brief Information; Drug: Cessation Phase Nicotine Patch + Nicotine Mini-Lozenge
- Reduction/Brief Info+Brief Info (Active Comparator): This arm includes Phase 2 (Preparation) Reduction Treatment and Phase 3 (Cessation) Brief Information. More specifically, treatments include the following:
  Phase 2: Nicotine Mini-Lozenge for 11 Months; Preparation Phase Behavioral Reduction Counseling;
  Phase 3: Cessation Phase Brief Information; Cessation Phase Nicotine Patch + Nicotine Mini-Lozenge
  Interventions: Drug: Nicotine Mini-Lozenge for 11 Months; Behavioral: Preparation Phase Behavioral Reduction Counseling; Behavioral: Cessation Phase Brief Information; Drug: Cessation Phase Nicotine Patch + Nicotine Mini-Lozenge
- Recycling/Supportive+Skill Counseling (Active Comparator): This arm includes Phase 2 (Preparation) Recycling Treatment and Phase 3 (Cessation) Supportive Counseling and Skill Training Counseling. More specifically, treatments include the following:
  Phase 2: Preparation Phase Recycling Counseling;
  Phase 3: Cessation Phase Supportive Counseling; Cessation Phase Skill Training Counseling; Cessation Phase Nicotine Patch + Nicotine Mini-Lozenge
  Interventions: Behavioral: Preparation Phase Recycling Counseling; Behavioral: Cessation Phase Supportive Counseling; Behavioral: Cessation Phase Skill Training Counseling; Drug: Cessation Phase Nicotine Patch + Nicotine Mini-Lozenge
- Recycling/Supportive Counsel+Brief Info (Active Comparator): This arm includes Phase 2 (Preparation) Recycling Treatment and Phase 3 (Cessation) Supportive Counseling and Brief Information. More specifically, treatments include the following:
  Phase 2: Preparation Phase Recycling Counseling;
  Phase 3: Cessation Phase Supportive Counseling; Cessation Phase Brief Information; Cessation Phase Nicotine Patch + Nicotine Mini-Lozenge
  Interventions: Behavioral: Preparation Phase Recycling Counseling; Behavioral: Cessation Phase Supportive Counseling; Behavioral: Cessation Phase Brief Information; Drug: Cessation Phase Nicotine Patch + Nicotine Mini-Lozenge
- Recycling/Skill Counsel+Brief Info (Active Comparator): This arm includes Phase 2 (Preparation) Recycling Treatment and Phase 3 (Cessation) Skill Training Counseling and Brief Information. More specifically, treatments include the following:
  Phase 2: Preparation Phase Recycling Counseling;
  Phase 3: Cessation Phase Skill Training Counseling; Cessation Phase Brief Information; Cessation Phase Nicotine Patch + Nicotine Mini-Lozenge
  Interventions: Behavioral: Preparation Phase Recycling Counseling; Behavioral: Cessation Phase Skill Training Counseling; Behavioral: Cessation Phase Brief Information; Drug: Cessation Phase Nicotine Patch + Nicotine Mini-Lozenge
- Recycling/Brief Info+Brief Info (Active Comparator): This arm includes Phase 2 (Preparation) Recycling Treatment and Phase 3 (Cessation) Brief Information. More specifically, treatments include the following:
  Phase 2: Preparation Phase Recycling Counseling;
  Phase 3: Cessation Phase Brief Information; Cessation Phase Nicotine Patch + Nicotine Mini-Lozenge
  Interventions: Behavioral: Preparation Phase Recycling Counseling; Behavioral: Cessation Phase Brief Information; Drug: Cessation Phase Nicotine Patch + Nicotine Mini-Lozenge
- Preparation Phase Control/No Phase 3 (Placebo Comparator): This arm includes Phase 2 (Preparation) Control Treatment and No Phase 3 (Cessation) Treatment. More specifically, treatments include the following:
  Phase 2: Preparation Phase Control Treatment
  Phase 3: No Treatment
  Interventions: Behavioral: Preparation Phase Control Treatment

INTERVENTIONS:
Drug: Nicotine Mini-Lozenge for 11 Months — Participants receive up to 11 months of Nicotine Mini-Lozenges as part of this treatment (dosing based on their nicotine dependence as measured when they started the study: 4 mg if they smoked within 30 minutes of waking and 2 mg if they smoked more than 30 minutes after waking, as per the package insert), along with instructions for use.
  Other Names: Nicotine Mini-Lozenge
  Arms: Reduction/Brief Info+Brief Info; Reduction/Skill Counseling+Brief Info; Reduction/Supportive Counsel+Brief Info; Reduction/Supportive+Skill Counseling
Behavioral: Preparation Phase Behavioral Reduction Counseling — Participants randomized to receive this treatment receive manual-based counseling calls and visits over the course of 11 months. The ultimate goal will be smoking that is reduced in amount and location. Case managers and participants will collaboratively identify a set of steps to progressively reduce smoking. The primary vehicles for change are to encourage substitution of the nicotine mini-lozenge for cigarettes and to reduce the contexts in which smoking occurs. Counseling will counter post-lapse demoralization by emphasizing participants' progress, the value of smoking reduction as a transitional goal, and the critical value of ongoing treatment engagement. Evidence of progress in reduction of smoking, and smoking contexts will be used to build self-efficacy.
  Other Names: Phase 2 Reduction Counseling
  Arms: Reduction/Brief Info+Brief Info; Reduction/Skill Counseling+Brief Info; Reduction/Supportive Counsel+Brief Info; Reduction/Supportive+Skill Counseling
Behavioral: Preparation Phase Recycling Counseling — Participants randomized to receive this treatment condition will be encouraged to commit to a new quit date as soon as they feel ready. In the counseling sessions, participants will be encouraged to discuss reasons for and concerns about quitting as well as barriers to setting a quit date.
  Other Names: Phase 2 Recycling Counseling
  Arms: Recycling/Brief Info+Brief Info; Recycling/Skill Counsel+Brief Info; Recycling/Supportive Counsel+Brief Info; Recycling/Supportive+Skill Counseling
Behavioral: Preparation Phase Control Treatment — Participants randomly assigned to the Preparation Phase Control Treatment condition will continue to receive the Initial Cessation usual care treatment (8 weeks of nicotine patch; two coaching sessions), but will also be told that they can receive additional treatment at no cost from the Wisconsin Tobacco Quitline (WTQL).
  Other Names: Phase 2 Control Treatment
  Arms: Preparation Phase Control/No Phase 3
Behavioral: Cessation Phase Supportive Counseling — Supportive Counseling will be consistent with the Public Health Service (PHS) Clinical Practice Guideline (Fiore et al., 2008) and will involve encouragement, a focus on short-term goals, discussion of participant values (what the participant feels would be good and healthy for them in the long run) and how these values are congruent with cessation, emphasis on the patient and the counselor being a team, encouragement for the participant to generate a quitting strategy with the message that smokers often have a good sense of what will work for them, and prompts for the participant to explore his/her feelings about quitting and feelings of optimism and concern (i.e., to use the counselor as a sounding board).
  Other Names: Phase 3 Supportive Counseling
  Arms: Recycling/Supportive Counsel+Brief Info; Recycling/Supportive+Skill Counseling; Reduction/Supportive Counsel+Brief Info; Reduction/Supportive+Skill Counseling
Behavioral: Cessation Phase Skill Training Counseling — Skill training Counseling will: 1) carefully assess smoking cue contexts and opportunities to smoke, to identify problems encountered in the prior quit attempt; 2) develop specific plans for avoiding such contexts and identify skills for coping with them; 3) develop plans for negotiating with others who smoke; 4) develop lifestyle changes to reduce future smoking opportunities and contexts; and 5) assign homework and assess execution of assigned skills. Participants will receive coping menus that provide personalized coping/avoidance options and "coping reports" that assess coping execution over time and troublesome contexts and cues around which counseling will be focused. There will be praise for any progress and a collaborative determination of barriers to skill execution.
  Other Names: Phase 3 Skill Training Counseling
  Arms: Recycling/Skill Counsel+Brief Info; Recycling/Supportive+Skill Counseling; Reduction/Skill Counseling+Brief Info; Reduction/Supportive+Skill Counseling
Behavioral: Cessation Phase Brief Information — Participants randomized to receive Brief Information will receive brief (generic) information about the importance of taking the cessation medication, how to use the medication, information about side effects/safety, and what to do in case of problems, and will also be given encouragement to quit smoking.
  Other Names: Phase 3 Brief Information
  Arms: Recycling/Brief Info+Brief Info; Recycling/Skill Counsel+Brief Info; Recycling/Supportive Counsel+Brief Info; Reduction/Brief Info+Brief Info; Reduction/Skill Counseling+Brief Info; Reduction/Supportive Counsel+Brief Info
Drug: Cessation Phase Nicotine Patch + Nicotine Mini-Lozenge — All participants will receive 8-weeks of combination NRT (nicotine patch + nicotine mini-lozenge). Nicotine patch dosing will be based on current cigarettes smoked per day, per package insert: for those who currently smoke >10 cigs/day=4 weeks of 21 mg, 2 weeks of 14 mg, and 2 weeks of 7 mg nicotine patches, along with nicotine mini-lozenges; for those who currently smoke <=10 cigs/day=6 weeks of 14 mg and 2 weeks of 7 mg nicotine patches along with mini-lozenges. Mini-lozenge dosing will be based on how soon participants currently smoke after waking before their initial quit attempt and will be consistent with the package insert (4 mg for participants who smoke within 30 minutes of waking and 2 mg for participants smoke more than 30 minutes after waking).
  Other Names: Cessation Phase Combination NRT
  Arms: Recycling/Brief Info+Brief Info; Recycling/Skill Counsel+Brief Info; Recycling/Supportive Counsel+Brief Info; Recycling/Supportive+Skill Counseling; Reduction/Brief Info+Brief Info; Reduction/Skill Counseling+Brief Info; Reduction/Supportive Counsel+Brief Info; Reduction/Supportive+Skill Counseling

SUMMARY:
Relapse after a serious quit attempt occurs in 70-90% of smokers who try to quit smoking. This study utilizes a sequential, multiple assignment, randomized trial (SMART) design - - an innovative multi-phase approach - - to test post-relapse treatments designed to assist smokers to make a new, successful quit attempt. This study will test Relapse Recovery (RR) treatments that are applied at two stages following relapse: 1) RR Preparation Phase treatments for smokers who relapse after an initial quit attempt, and 2) RR Cessation Phase treatments for relapsed smokers who decide to make a new quit attempt. Smokers motivated to quit smoking will make an initial quit attempt in the Quit Phase (cessation medication + counseling). Participants who relapse will be randomized to one of three RR Preparation Phase treatments (Behavioral [Smoking] Reduction Counseling + the Nicotine Mini-Lozenge; Recycling Counseling that encourages participants to quit again as soon as possible; and Preparation Phase Control). RR Preparation Phase participants (other than controls) who elect to try a new quit attempt will be randomized to one of four RR Cessation Phase treatments based on a 2X2 fully-crossed factorial design testing two factors: Supportive Counseling (vs. Brief Information) and Skill Training (vs. Brief Information). All RR Cessation Phase participants will receive 8 weeks of combination nicotine replacement therapy (nicotine patch + nicotine mini-lozenge). The investigators hypothesize that RR Preparation Phase Reduction treatment will significantly increase long-term abstinence rates relative to the Preparation Phase Control condition.

DETAILED DESCRIPTION:
This study aims to identify effective Relapse Recovery (RR) treatments to assist smokers who relapse after an initial quit attempt. The study will use a sequential, multiple assignment, randomized trial (SMART) design with three phases. In a SMART design, randomization occurs at more than one stage, with randomization at a later stage based on response to treatment at an earlier stage. The three phases in this SMART study are as follows:

1. Phase 1 consists of the Quit Phase in which all participants (smokers motivated to quit smoking) will be offered evidence-based cessation treatment (cessation medication plus counseling). Participants who relapse will be eligible to proceed to the next phase which involves Relapse Recovery (RR) Preparation treatment.
2. Phase 2 consists of RR Preparation Phase treatments in which relapsed participants from the Quit Phase will be randomized to three arms: (a) Recycling Counseling (where participants are encouraged to quit again as soon as possible); (b) Behavioral Reduction Counseling + Nicotine Mini-Lozenge (which targets smoking reduction and preparation for a new quit attempt); and (c) Preparation Phase Control (continuation of Quit Phase treatment plus advice to seek additional help from the Wisconsin Tobacco Quit Line or their clinic care provider).
3. Phase 3 consists of RR Cessation Phase treatments in which non-control (i.e. Recycling or Behavioral Reduction) Preparation Phase participants who elect to make a new quit attempt will be randomized to one of four treatment conditions in a 2X2 fully-crossed factorial design: (a) Supportive Counseling + Skill Training; (b) Supportive Counseling + Brief Information; (c) Skill Training + Brief Information; and (d) Brief Information Only. All participants will receive 8 weeks of combination nicotine replacement therapy (Nicotine Patch + Nicotine Mini-Lozenge). Brief Information will consist of generic information about the importance of taking the medication and how to use it, information about side effects/safety and what to do in case of problems, and participants will also be given encouragement.

Smoking status will be assessed 14 months after randomization to RR Preparation Phase treatment. The investigators hypothesize that 7-day point point-prevalence abstinence rates will be 15% for the Preparation Phase Control condition, 25% for the Recycling condition, and 35% for the Behavioral Reduction condition. The investigators propose that any increase in abstinence of 15% or higher would be clinically significant. The investigators did not power the study to demonstrate a significant difference between the two active RR Preparation Phase treatments. Therefore, the investigators anticipate that only the RR Behavioral Reduction treatment will significantly increase long-term abstinence rates (primary outcome: Biochemically-confirmed 7-Day Point Prevalence Abstinence at 14 Months post-randomization to Phase 2 Preparation treatment) over those produced by the Preparation Phase Control condition. Because of limitations in statistical power, analyses of RR Cessation Phase treatments will be exploratory only (secondary outcome: Self-Reported 7-Day Point Prevalence Abstinence at 26 Weeks post-randomization to Phase 3 Cessation treatment).

ELIGIBILITY:
Inclusion Criteria:

1. age >=18 years,
2. smoking >4 cigarettes/day for the previous 6 months,
3. able to read, write, and speak English,
4. have reliable phone access and agree to respond to Interactive Voice Response (IVR) phone prompts, and
5. if currently using NRT, agreeing to use only study medication for the duration of the study, we will not exclude participants based on their prior use of cessation medication or if they use multiple tobacco products in order to enhance real-world generalization (these will be statistically controlled in analyses),
6. motivation to quit smoking, and
7. planning to remain in the intervention catchment area for at least 2 years and 2 months, .

Exclusion Criteria:

1. Currently taking bupropion or varenicline,
2. unwillingness to cease other forms of nicotine replacement or Chantix (also called Varenicline),
3. medical contraindications to using NRT including hospitalized (for at least one night) for a stroke, heart attack, congestive heart failure or diabetes in the last 4 weeks, history of a serious skin or allergic reaction to using the Nicotine patch,
4. diagnosis of or treatment for schizophrenia, a psychotic disorder or bipolar disorder in the last 10 years and,
5. if the participant is a woman of childbearing potential, being pregnant or intending to becoming pregnant or unwillingness to use an approved method of birth control during treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1154 (Actual)
Dates: Start 2015-10-30 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Biochemically-confirmed 7-Day Point Prevalence Abstinence | 14 Months after randomization to Phase 2 Preparation treatment
  Participants who self-report no smoking for the past 7 days at the assessment endpoint (14 months post-randomization to Phase 2 Preparation treatment) and who provide an exhaled breath sample for carbon monoxide testing with a concentration no higher than 5 parts per million will be considered to meet criteria for Biochemically-confirmed 7-Day Point Prevalence Abstinence. Participants who do not meet these criteria will be considered to be relapsed (smoking).

SECONDARY OUTCOMES:
Self-Reported 7-Day Point Prevalence Abstinence | 26 Weeks after randomization to the Phase 3 Cessation treatment
  Participants who self-report no smoking for the past 7 days at the assessment endpoint (26 weeks post-randomization to Phase 3 Cessation treatment) will be considered to meet criteria for Self-Reported 7-Day Point Prevalence Abstinence. Participants who report any smoking in the past 7 days at the assessment endpoint will be considered to be relapsed (smoking).

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Schlam, PhD, Study Director — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Center for Tobacco Research and Intervention, School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make the final de-identifed datasets available in standard file formats by request from other researchers in a timely manner (no later than the acceptance for publication of the main findings from the final dataset).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After publication of the main findings.
Access Criteria: Approval of a data request by the investigators.

REFERENCES:
- [Derived] Schlam TR, Baker TB, Piper ME, Cook JW, Smith SS, Zwaga D, Jorenby DE, Almirall D, Bolt DM, Collins LM, Mermelstein R, Fiore MC. What to do after smoking relapse? A sequential multiple assignment randomized trial of chronic care smoking treatments. Addiction. 2024 May;119(5):898-914. doi: 10.1111/add.16428. Epub 2024 Jan 28. PMID 38282258
- See also: University of Wisconsin Center for Tobacco Research and Intervention — http://www.ctri.wisc.edu/